CLINICAL TRIAL: NCT04209608
Title: Observational Study on Respiratory Impact of High-frequency Jet Ventilation (JVHF) in Interventional Radiology (RI)
Acronym: Pulmojet
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC19_0416
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Anesthesia Complication

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Jet ventilation is used in interventional radiology to reduce respiratory movement and facilitate tumor destruction. The purpose of this study is to describe the respiratory impact of this technique

DETAILED DESCRIPTION:
Use imaging and respiratory data to describe the impact of JVHF during tumor thermoablation procedures

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Patient benefiting from an abdominal tumor thermoablation procedures
* Patient who gave consent
* Patient with a social protection scheme

Exclusion Criteria:

* Pulmonary thermoablation procedures
* Thermoablation of abdominal tumors required a transpleural passage
* Patient under guardianship or curatorship
* Patient not understanding French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be offered to patients benefiting from thermoablation of abdominal tumors under JVHF. Recruitment will take place during the pre-anesthetic consultation.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
evaluate the respiratory impact after the use of JVHF after thermoablation of a solid abdominal tumour. | through study completion, an average of 1 year
  Respiratory complication rate.

SECONDARY OUTCOMES:
Describe the number of ventilatory disorders | through study completion, an average of 1 year
  Score Radiological Atelectasis Score (RAS) of Richter Larsen - RAS: 0, clear lung field; 1, plate like atelectasis or slight infiltration; 2, partial atelectasis; 3, lobar atelectasis; 4, bilateral lobar atelectasis.
Describe the incidence of hypoxemia during JVHF | through study completion, an average of 1 year
  Difference between oxygen saturation at the end of the procedure and at the beginning of the procedure
Describe the incidence of hypercapnia at the time of a JVHF | through study completion, an average of 1 year
  Difference between end of procedure and beginning of procedure capnia
Describe the incidence of barotraumatic pulmonary lesions at the time of a JVHF | through study completion, an average of 1 year
  Presence of barotraumatic pulmonary lesions on the imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trochu T, Desfriches-Doria N, Grillot N, Feuillet F, Lair D, Liberge R, Douane F, Dumont R, David A. Safety of High-Frequency Jet Ventilation During Image-Guided Thermal Ablation Procedures. Cardiovasc Intervent Radiol. 2023 Mar;46(3):360-368. doi: 10.1007/s00270-023-03358-5. Epub 2023 Jan 19. PMID 36658374